CLINICAL TRIAL: NCT05743959
Title: ctDNA Detection of MRD in Predicting Postoperative Recurrence in Biliary Tract Cancers：A Multicenter Prospective Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Dominant_2022
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Biliary Tract Cancer
Keywords: Cholangiocarcinoma; ctDNA; Minimal Residual Disease (MRD)
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stage I-III biliary tract cancers: Patients with stage I-III biliary tract cancers eligible for curative surgical resection
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: No intervention — No intervention

SUMMARY:
A substantial proporation of patients with biliary tract malignancies still experience disease recurrence after curative resection. ctDNA-based minimal residual disease (MRD) method has been widely used to monitor postoperative recurrence in solid cancers, but few studies have been reported in biliary tract cancers.

The present clinical trial aims to elucidate the correlation between the postoperative ctDNA status and the prognosis of patients with biliary tract cancers, and evaluate whether ctDNA could better predict patients' recurrence and guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age on the day of signing informed consent.
2. Clinically diagnosed as BTC before surgery and confirmed by pathology after surgery.
3. Stage I-III tumor according to the UICC/AJCC TNM staging system (8th edition in 2017), meeting the indications for radical surgery and are planned to undergo radical treatment. Those who do not undergo radical surgery will be excluded.
4. Patients must have a performance status of ≤1 on the ECOG Performance Scale.
5. Patients must have survival of > 6 months after surgery
6. Serological tumor indicators (CEA, CA19-9) and imaging data ( CT and/or MRI, PET-CT) were complete.
7. Blood biochemical indicators meet surgical standards
8. Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

1. Patients with recurrent biliary tract tumors
2. Patients with hepatobiliary mixed tumors
3. Patients with malignant tumors of other organs that have not been cured before.
4. History of organ transplant or allogeneic stem cell transplant
5. Patients with severe infections that are active or poorly controlled clinically
6. patients who are cognitively impaired or with known psychiatric disorders, and/or substance abuse
7. pregnant or lactating women
8. Failed to sign informed consent
9. Other conditions that researchers judged inappropriate for inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III biliary duct cancer eligible for curative surgical resection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | through study completion, an average of 2 years
  The primary endpoint for this study is Relapse-free survival (RFS), which will be assessed using RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcheng Li, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with NanJing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No